CLINICAL TRIAL: NCT06718452
Title: Treatment of Tinnitus Targeting Neuroinflammation. umPEALUT as Possible Option
Brief Title: Tinnitus and Treatment With umPEA-LUT
Acronym: TiniPEA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: Universita degli Studi di Napoli Federico (Unknown)
Responsible Party: Principal Investigator, Arianna Di Stadio, Associate Professor definite time, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UniLINK2026; University LINK (Other: Public Institution)
Record Dates: First submitted 2024-11-28; First posted 2024-12-05 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Tinnitus; Neuroinflammation
Keywords: Tinnitus; Neuroinflammation; Palmitoyetanolamide; Luteolin; Ultramicronized; Vascular; Central; Peripheral; Auditory cortex; Inner ear
MeSH Terms: conditions — Tinnitus; Neuroinflammatory Diseases | interventions — Rutin; 5-Hydroxytryptophan

STUDY DESIGN:
Intervention Model Description: Longitudinal study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Patients in this group will be treated using placebo
  Interventions: Dietary Supplement: Placebo
- Ultramicronized PEALUT Double dose (Experimental): umPEALUT 2 sachet/day every day for 60 days
  Interventions: Dietary Supplement: PEA-LUT 2 sachet day
- TREATMENT 2 (Experimental): umPEALUT 2 sachets day + 120 mg Rutin +100 mg 5 hTp
  Interventions: Combination Product: umPEALUT + Rutin + 5 hTp

INTERVENTIONS:
Dietary Supplement: PEA-LUT 2 sachet day — 1 sachet two times a day to be sublingually absorbed
  Arms: Ultramicronized PEALUT Double dose
Dietary Supplement: Placebo — Same administration of PEA-LUT
  Arms: Placebo
Combination Product: umPEALUT + Rutin + 5 hTp — People in this group will be treated by 2 sachets par day of umPEALUT associated to 120 mg of rutin and 100 mg of 5 hTp
  Arms: TREATMENT 2

SUMMARY:
Tinnitus can have different causes. From a peripheral point of view, the sensation of hearing a not present sound can be indicative of damage in the cells of the cochlea. Damage at this level can arise from traumatic, vascular, toxic origins or be caused by systemic pathologies. However, all the previous causes have a common denominator, the presence of reactive oxygen species (ROS), in the cochlea which determines the damage and the consequent death of the hair cells into the ear. The sound (tinnitus) that the patient perceives is generated by the spontaneous movement of the cilia of the hair cells; this phenomenon arises when these cells begin to be damaged.

Tinnitus can be also caused by a retrocochlear disorder such as damage of the auditory nerve (inflammatory and tumor cause). In case of an inflammatory origin, the factors released during inflammation can locally damage the nerves and spread into the cochlea destroying the hair cells.

Tinnitus can also originate from damage in the central auditory pathway. In this case, the problem persistent. It is important to keep in mind that although initially the tinnitus may originate from a damage inside the cochlea, after 6 months of persistence chronicizes causing an activation (without stimulus) of the upper auditory areas. This zone of "hypersensitivity" is therefore responsible for chronic tinnitus.

In addition to the overmentioned medical causes, tinnitus can also be sign of psychiatric/psychological disorders, in those cases in whom there is an involvement of the hypothalamus, as showed by neuropsychological studies. Tinnitus can be temporary and disappear spontaneously or, in the most of cases, be persistent and extremely annoying/stressful for the patient. At night in particular, in the absence of noise, the patient suffers more the presence of this ghost sound, which in some occasions prevents sleep. Insomnia negatively impacts on tinnitus increasing its duration and intensity, thus establishing a perpetual cycle of stress into the brain. The latter phenomenon worses and chronicizes the symptom .

Stress causes inflammation with ROS increase, which can affect both the peripheral and central auditory pathways. Recently, it has been shown that tinnitus can be a symptom of neuro-inflammatory pathologies such as, for example, Multiple Sclerosis.

The effects of inflammation on the hair cells are identifiable only through electrophysiological studies or from the temporal bone.

Keeping on mind inflammation and neuro-inflammation and considering the exchange between cerebrospinal fluid and perilymph , we speculate that the use of a molecule capable of reducing inflammation and modulating the action of mast cells and microglia, could be an effective tool to resolve tinnitus; moreover, thanks to its powerful action at the level of neuro-inflammation, it could reduce the hyper-activity in the upper auditory tracts, thus reducing/abolishing noise.

umPeaLut combines palmitoylethanolamide, which modulates the activity of mast cells, macrophages and microglia and luteolin, a bioflanoid extracted from fruits with anti-oxidant properties, able to improve microcirculation. Because the alterations of the ear microcirculation can be an additional cause of tinnitus, we believe that luteolin content can be an ulterior benefit.

Although various attempts have been made to use a mono-molecule, recent studies have shown that combination of several elements could reduce tinnitus ; PeaLut, in its ultra-micronized form with high bioavailability, could be the perfect solution.

This study aims at evaluating the efficacy of umPEALUT as a therapeutic treatment of tinnitus in a sample of adults.

DETAILED DESCRIPTION:
Longitudinal study on 100 patients

Patients between 18 and 70 years of age, not affected by systemic disorders (hypertension, diabetes, neurological disorders, previous stroke) or known psychological/psychiatric disorders will be included.

The patients will be evaluated at three observation times: T0 before treatment at the time of enrollment, T3 after 3 months and T6 after six months of treatment.

All patients, at each check-point will be screened as following: 1) three questionnaire to evaluate Tinnitus and 2) audiometric examination and acuphenometry.

Patients will be randomized into three groups, one group (CONTROL) that will use placebo, one (TREATMENT1 ) group that will use umPEALUT 2 sachets for day, and the other group (TREATMENT 2) umPEALUT 2 sachets par day combined to 120 mg of Rutin and 100 of 5-hTP.

EXPECTED RESULTS

Patients treated with umPEALUT compared to the control group will present an improvement of the symptom due to the anti-ROS action of luteolin and the neuro-immuno-modulating action of PEA. However the combination of umPEALUt with rutin and 5hTp will have better results than treatment with umPEALUT alone and control.

The changes induced by the treatment will be identifiable through the improvement of the symptom (responses to the questionnaire) and the changes in the subjective auditory test.

Specifically, patients in group 1 will present better final values than group 2, although group 2 will, however, present improvements compared to the control.

ELIGIBILITY:
Inclusion Criteria:

- Patients with tinnitus not under treatment at least for 30 days

Exclusion Criteria:

* Stroke in the last year
* Uncontrolled diabetes,
* Uncontrolled hypertension,
* Severe psychiatric disorders,
* Severe cognitive decline,
* Previous surgery of the brain or audio-vestibular nerves

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-04-20 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Tinnitus | At Enrollement, after 3 months of treatment, after 6 months of treatment (end of the therapy)
  Tinnitus questionnaire

SECONDARY OUTCOMES:
Auditory test | Enrollement (T0) and after 6 months (end of the therapy)
  Pure Tone Auditory test

CONTACTS AND LOCATIONS:
Overall Officials: Arianna Di Stadio, MD, PhD, MSc, Study Chair — Vanvitelli University
Locations (1):
- Vanvitelli ENT department, Naples, Campania, Italy

IPD SHARING:
Plan to Share IPD: Undecided
We are thinking about put everything in a repository

REFERENCES:
- [Result] Polanski JF, Soares AD, de Mendonca Cruz OL. Antioxidant therapy in the elderly with tinnitus. Braz J Otorhinolaryngol. 2016 May-Jun;82(3):269-74. doi: 10.1016/j.bjorl.2015.04.016. Epub 2015 Oct 17. PMID 26547700
- [Result] Petridou AI, Zagora ET, Petridis P, Korres GS, Gazouli M, Xenelis I, Kyrodimos E, Kontothanasi G, Kaliora AC. The Effect of Antioxidant Supplementation in Patients with Tinnitus and Normal Hearing or Hearing Loss: A Randomized, Double-Blind, Placebo Controlled Trial. Nutrients. 2019 Dec 12;11(12):3037. doi: 10.3390/nu11123037. PMID 31842394
- [Result] Wicinski M, Socha M, Walczak M, Wodkiewicz E, Malinowski B, Rewerski S, Gorski K, Pawlak-Osinska K. Beneficial Effects of Resveratrol Administration-Focus on Potential Biochemical Mechanisms in Cardiovascular Conditions. Nutrients. 2018 Nov 21;10(11):1813. doi: 10.3390/nu10111813. PMID 30469326
- [Result] Facchinetti R, Valenza M, Bronzuoli MR, Menegoni G, Ratano P, Steardo L, Campolongo P, Scuderi C. Looking for a Treatment for the Early Stage of Alzheimer's Disease: Preclinical Evidence with Co-Ultramicronized Palmitoylethanolamide and Luteolin. Int J Mol Sci. 2020 May 27;21(11):3802. doi: 10.3390/ijms21113802. PMID 32471239
- [Result] Di Stadio A, Ralli M. Inner ear involvement in multiple sclerosis: An underestimated condition? Mult Scler. 2018 Aug;24(9):1264-1265. doi: 10.1177/1352458517750010. No abstract available. PMID 30015600
- [Result] Albanese M, Di Girolamo S, Silvani L, Ciaschi E, Chiaramonte B, Conti M, Passali FM, Di Gioia B, Mercuri NB, Di Stadio A. Distortion Product Otoacoustic Emissions and Their Suppression as Predictors of Peripheral Auditory Damage in Migraine: A Case-Control Study. J Clin Med. 2021 Oct 27;10(21):5007. doi: 10.3390/jcm10215007. PMID 34768526
- [Result] Cronlein T, Langguth B, Geisler P, Hajak G. Tinnitus and insomnia. Prog Brain Res. 2007;166:227-33. doi: 10.1016/S0079-6123(07)66021-X. PMID 17956787
- [Result] Mazurek B, Szczepek AJ, Hebert S. Stress and tinnitus. HNO. 2015 Apr;63(4):258-65. doi: 10.1007/s00106-014-2973-7. PMID 25862619
- [Result] Xu Y, Shi Y, Yao J, Yang H, Ding Z, Chen QQ, Liu Y, Chen W. Altered brain functional connectivity and correlation with psychological status in patients with unilateral pulsatile tinnitus. Neurosci Lett. 2019 Jul 13;705:235-245. doi: 10.1016/j.neulet.2019.04.046. Epub 2019 Apr 28. PMID 31042571
- [Result] Andersson G. Psychological aspects of tinnitus and the application of cognitive-behavioral therapy. Clin Psychol Rev. 2002 Sep;22(7):977-90. doi: 10.1016/s0272-7358(01)00124-6. PMID 12238249
- [Result] Shulman A, Wang W, Luo H, Bao S, Searchfield G, Zhang J. Neuroinflammation and Tinnitus. Curr Top Behav Neurosci. 2021;51:161-174. doi: 10.1007/7854_2021_238. PMID 34282564
- [Result] Galazyuk AV, Wenstrup JJ, Hamid MA. Tinnitus and underlying brain mechanisms. Curr Opin Otolaryngol Head Neck Surg. 2012 Oct;20(5):409-15. doi: 10.1097/MOO.0b013e3283577b81. PMID 22931904
- [Result] Savastano M, Brescia G, Marioni G. Antioxidant therapy in idiopathic tinnitus: preliminary outcomes. Arch Med Res. 2007 May;38(4):456-9. doi: 10.1016/j.arcmed.2006.12.004. Epub 2007 Mar 12. PMID 17416295
- [Result] Naunton RF, Proctor L, Elpern BS. The audiologic signs of ninth nerve neurinoma. Arch Otolaryngol. 1968 Mar;87(3):222-7. doi: 10.1001/archotol.1968.00760060224002. No abstract available. PMID 5642369
- [Result] Di Stadio A, Dipietro L, Ralli M, Meneghello F, Minni A, Greco A, Stabile MR, Bernitsas E. Sudden hearing loss as an early detector of multiple sclerosis: a systematic review. Eur Rev Med Pharmacol Sci. 2018 Jul;22(14):4611-4624. doi: 10.26355/eurrev_201807_15520. PMID 30058696
- [Result] Norena AJ. Revisiting the cochlear and central mechanisms of tinnitus and therapeutic approaches. Audiol Neurootol. 2015;20 Suppl 1:53-9. doi: 10.1159/000380749. Epub 2015 May 19. PMID 25997584
- [Result] Lechtenberg R, Shulman A. The neurologic implications of tinnitus. Arch Neurol. 1984 Jul;41(7):718-21. doi: 10.1001/archneur.1984.04050180040014. PMID 6743061
- [Result] Samlan SR, Jordan MT, Chan SB, Wahl MS, Rubin RL. Tinnitus as a measure of salicylate toxicity in the overdose setting. West J Emerg Med. 2008 Aug;9(3):146-9. PMID 19561730
- [Result] Figueiredo RR, de Azevedo AA, Penido Nde O. Tinnitus and arterial hypertension: a systematic review. Eur Arch Otorhinolaryngol. 2015 Nov;272(11):3089-94. doi: 10.1007/s00405-014-3277-y. Epub 2014 Sep 5. PMID 25190255
- [Result] Ralli M, Balla MP, Greco A, Altissimi G, Ricci P, Turchetta R, de Virgilio A, de Vincentiis M, Ricci S, Cianfrone G. Work-Related Noise Exposure in a Cohort of Patients with Chronic Tinnitus: Analysis of Demographic and Audiological Characteristics. Int J Environ Res Public Health. 2017 Sep 8;14(9):1035. doi: 10.3390/ijerph14091035. PMID 28885581
- [Result] Di Stadio A, Dipietro L, Ricci G, Della Volpe A, Minni A, Greco A, de Vincentiis M, Ralli M. Hearing Loss, Tinnitus, Hyperacusis, and Diplacusis in Professional Musicians: A Systematic Review. Int J Environ Res Public Health. 2018 Sep 26;15(10):2120. doi: 10.3390/ijerph15102120. PMID 30261653
- [Result] Haider HF, Bojic T, Ribeiro SF, Paco J, Hall DA, Szczepek AJ. Pathophysiology of Subjective Tinnitus: Triggers and Maintenance. Front Neurosci. 2018 Nov 27;12:866. doi: 10.3389/fnins.2018.00866. eCollection 2018. PMID 30538616